CLINICAL TRIAL: NCT00772902
Title: A Phase 4, Open Label, Randomized, Controlled Study to Assess the Effect on Lipid Profile of Switching a Stable HAART Regimen of Fixed Dose Abacavir/Lamivudine (Kivexa) Plus Lopinavir/Ritonavir (Kaletra), to Emtricitabine/Tenofovir Disoproxil Fumarate (Truvada) Plus Lopinavir/Ritonavir (Kaletra) in Adult HIV-1 Infected Subjects With Raised Cholesterol
Brief Title: ROCKET II - Randomized Open Label Switch for Cholesterol Elevation on Kivexa + Kaletra Evaluation Trial
Acronym: ROCKET II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-EU-164-0206; 2008-002043-16 (EudraCT Number)
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: HIV-1
Keywords: HIV-1; LDL; HDL; non-HDL cholesterol; triglycerides; cholesterol
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; lopinavir-ritonavir drug combination; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Truvada + Kaletra (Experimental): Truvada (emtricitabine 200 mg/tenofovir DF 300 mg) once daily for oral administration according to prescription information. As third agent, continuing Kaletra (lopinavir 200 mg/ritonavir 50 mg) for oral administration according to prescription.
  Interventions: Drug: Truvada + Kaletra
- Kivexa + Kaletra (Active Comparator): Continuing Kivexa (abacavir sulfate 600 mg/lamivudine 300 mg) once daily for oral administration according to prescription. As third agent, continuing Kaletra (lopinavir 200 mg/ritonavir 50 mg) for oral administration according to prescription.
  Interventions: Drug: Kivexa + Kaletra

INTERVENTIONS:
Drug: Truvada + Kaletra — Truvada (emtricitabine 200 mg/tenofovir DF 300 mg)once daily for oral administration according to prescription information. As third agent, continuing Kaletra (lopinavir 200 mg/ritonavir 50 mg) for oral administration according to prescription.
  Arms: Truvada + Kaletra
Drug: Kivexa + Kaletra — Continuing Kivexa (abacavir sulfate 600 mg/lamivudine 300 mg) once daily for oral administration according to prescription. As third agent, continuing Kaletra (lopinavir 200 mg/ritonavir 50 mg) for oral administration according to prescription.
  Other Names: Kivexa = Epzicom
  Arms: Kivexa + Kaletra

SUMMARY:
This study investigated whether human immunodeficiency virus type 1 (HIV-1) infected subjects with raised cholesterol switching their nucleoside reverse transcriptase inhibitor (NRTI) backbone from Kivexa (Epzicom) to Truvada had an improvement in their fasting total cholesterol after 12 weeks of treatment. The study also investigated whether any improvement had a beneficial effect on the overall cardiovascular risk.

DETAILED DESCRIPTION:
This was a Phase 4, open-label, randomized, multicenter (in the European Union), controlled study to assess the effect on lipid profile of switching from a stable highly active antiretroviral therapy (HAART) regimen of Kivexa + Kaletra to Truvada + Kaletra in adult HIV-1 infected subjects with raised cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Plasma HIV-1 RNA < 50 copies/mL at screening and for ≥ 12 weeks prior to Screening
* Stable HAART regimen of Kivexa + Kaletra for ≥ 24 weeks prior to Screening
* Documented confirmed raised total cholesterol ≥ 5.2 mmol/L (≥ 200 mg/dL) for the last two consecutive tests (at least 4 weeks apart)
* Fasted total cholesterol ≥ 5.2 mmol/L (≥ 200 mg/dL) at Screening
* Subject willing to continue current unmodified HAART for 12 weeks if randomized to Group 2
* Subjects requiring concomitant lipid regulating therapy must be established on a stable dose/frequency ≥ 12 weeks prior to Screening and be expected to remain stable in dose and frequency throughout the treatment phase of the study. Simvastatin and lovastatin are not allowed.
* Adequate renal function by calculated creatinine clearance ≥ 60 mL/min according to the Cockcroft-Gault formula
* Negative serum pregnancy test (females of childbearing potential only i.e., not surgically sterile or at least 2 years post-menopausal)
* Serum Total Bilirubin ≤ 1.5 mg/dL (Note: In cases of clinically insignificant, asymptomatic elevated Serum Total Bilirubin [e.g. due to Gilbert Syndrome] the subject may be enrolled in the study with Serum Total Bilirubin >1.5 mg/dL with the agreement of the Medical Monitor)
* Women of childbearing potential (WOCBP) must be using a highly effective method of contraception to avoid pregnancy throughout the study and for up to 30 days after the last dose of study drugs in such a manner that the risk of pregnancy is minimized
* Female subjects who are postmenopausal for less than 2 years are required to have follicle stimulating hormone (FSH) ≥ 40 mIU/mL. If the FSH is < 40 mIU/mL, the subject must agree to use highly effective method of birth control to participate in the study.
* Male subjects who are sexually active must be willing to use effective barrier contraception (e.g. condom with spermicide) during heterosexual intercourse from screening through completion of the study and continuing for up to 30 days after the last dose of study drugs
* Life expectancy ≥ 1 year
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.

Exclusion Criteria:

* Pregnant or lactating subjects
* Previous treatment with emtricitabine (FTC), tenofovir DF (TDF) or adefovir dipivoxil (ADV)
* Known hypersensitivity to emtricitabine (FTC), tenofovir DF (TDF), Truvada or any of the excipients (e.g., lactose monohydrate)
* Documented resistance to any of the study drugs (either genotypic or phenotypic)
* Severe hepatic impairment
* Hepatitis B infection with viral load > 1000 copies/mL at Screening or Hepatitis C infection requiring therapy
* Treatment with any interferon or pegylated interferon within 18 months prior to Screening
* Hepatic transaminases (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) ≥ 5 × upper limit of normal (ULN)
* Subjects receiving ongoing therapy with any of the medications that are contraindicated with any of the study drugs. Administration of any of these medications must be discontinued at least 28 days prior to the Baseline visit and for the duration of the study period.
* Active, serious infections (other than HIV infection) requiring parenteral antibiotic therapy within 15 days prior to screening
* Prior history of significant renal or bone disease
* Any current known clinical or symptomatic laboratory parameter of Gilead Sciences, Inc., Grade 4. Asymptomatic Grade 4 abnormalities will be permitted at the discretion of the investigator if deemed clinically appropriate (excluding adverse events and laboratory parameters mentioned elsewhere in the inclusion/exclusion criteria). Abnormalities deemed insignificant by the investigator must be discussed with the Medical Monitor prior to enrollment.
* Malignancy other than cutaneous Kaposi sarcoma (KS) or basal cell carcinoma. Subjects with biopsy-confirmed cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of baseline and are not anticipated to require systemic therapy during the study
* Current alcohol or substance use judged by the investigator to potentially interfere with subject study compliance
* Subjects currently taking part in any other clinical trial using an investigational product, with the exception of studies where the treatment studied has been stopped for more than 1 month prior to baseline
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine if switching the NRTI backbone from Kivexa to Truvada leads to a reduction in fasting total cholesterol at 12 weeks. | 12 weeks

SECONDARY OUTCOMES:
Evaluation of fasting metabolic parameters (e.g. LDL, HDL, non-HDL cholesterol, triglycerides and cholesterol ratios). | 12 weeks
Evaluation of efficacy and safety by assessing adverse events, clinical laboratory tests, physical examinations and vital signs at every visit. | Upto 12 weeks
Evaluation of changes in the 10-year risk factor for coronary heart disease outcomes as measured by total cholesterol, HDL, blood pressure, smoking status, treatment for hypertension, sex, and age. | 10 year risk factor from 12 week evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Florian Abel, Study Director — Gilead Sciences
Locations (4):
- Gilead Sciences, Vienna, Austria
- Gilead Sciences, Munich, Germany
- Gilead Sciences, Milan, Italy
- Gilead Sciences, Madrid, Spain

REFERENCES:
- [Derived] Behrens G, Maserati R, Rieger A, Domingo P, Abel F, Wang H, Pearce G. Switching to tenofovir/emtricitabine from abacavir/lamivudine in HIV-infected adults with raised cholesterol: effect on lipid profiles. Antivir Ther. 2012;17(6):1011-20. doi: 10.3851/IMP2305. Epub 2012 Aug 15. PMID 22910324